CLINICAL TRIAL: NCT06460753
Title: Analysis of Laboratory Markers for Severe COVID-19
Status: Completed | Type: Observational
Sponsor: Karaganda Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SC19MI-ARICU-1T
Record Dates: First submitted 2024-06-12; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Coronavirus Infection COVID-19
Keywords: coronavirus infection; COVID-19; biochemical markers; forecasting; outcomes; resuscitation and intensive care
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — biochemical parameters: procalcitonin, C-reactive protein, D-dimer, ferritin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospitalized to ICU severe patients with coronavirus infection COVID-19: an analysis of the medical records was carried out
  Interventions: Diagnostic Test: CT of the chest organs, blood biochemical parameters

INTERVENTIONS:
Diagnostic Test: CT of the chest organs, blood biochemical parameters — Taking into account the clinical manifestations, all patients underwent chest computed tomography (CT) to diagnose COVID-19-associated pneumonia. According to the CT results, all patients were classified into one of 4 subgroups, according to the degree of pulmonary infiltration. The following biochemical parameters were selected and used to monitor dynamics: procalcitonin (PCT), C-reactive protein (CRP), D-dimer (DD), ferritin (FRT). Biochemical markers were determined daily during the stay in the intensive care unit. The duration of observation was 15 days was selected. Information was analysed retrospectively.

SUMMARY:
The course of coronavirus infection was often severe and required hospitalization of patients in the intensive care unit. The new SARS-Cov-2 has been poor studied, so relatively reliable markers are needed to effectively monitor patients and predict complications and outcome. Taking into account the known mechanisms of pathogenesis, the biochemical markers as ferritin, procalcitonin, C-reactive protein and D-dimer were chosen for this purpose. Patients were divided according to the degree of pulmonary infiltration. We hypothesized that the markers would correlate with dynamics, complications, and outcomes.

DETAILED DESCRIPTION:
In the presented study, an analysis of the medical records of 193 patients hospitalized in severe condition to the intensive care unit with a confirmed diagnosis of Coronavirus infection COVID-19 was carried out. Taking into account the volume of pulmonary infiltration according to computer tomography (CT) of the chest organs, patients were divided into 4 groups in accordance with the approved classification: CT 1(up to 25% of lung tissue was infiltrated) - 27 patients, CT 2 (25-50%) - 60 patients, CT 3 (50-75%) - 67 patients, CT 4 (75% and more) - 39 patients. The following biochemical parameters were selected and used to monitor dynamics: procalcitonin (PCT), C-reactive protein (CRP), D-dimer (DD), ferritin (FRT). The duration of observation was 15 days.

In order to determine correlations between quantitative and qualitative data at different stages of treatment, a correlation analysis was carried out (Spearman's test was used). ROC analysis was performed to evaluate selected laboratory markers as predictors of outcome. Next, the odds ratio (OR) was assessed taking into account the obtained Youden's J index and the Associated criterion for each of the selected markers in relation to the patient's outcome. Preliminary contingency tables were compiled in relation to laboratory parameters and outcomes (2x2 tables).

Data were processed using statistical software jamovi (Computer Software ,Version 2.3.26), MedCalc (MedCalc Software Ltd, Ostend, Belgium), Microsoft Office Excel, 2016.

ELIGIBILITY:
Inclusion Criteria:

* identified COVID-19 by nasopharyngeal material PCR, coronavirus associated lung infiltration, visualized by CT, and clinically severe condition

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the intensive care unit of the Regional Clinical Hospital of Karaganda, which is the clinical base of the Karaganda Medical University.
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Biochemical markers' correlation with outcomes | Laboratory markers were measured daily. For correlation analysis, control days of measurements were chosen: days 1-3-7-15.
  In the early stages of hospitalization was found the significant inverse correlation (p < 0.01, r -0.236) with the outcome of the stay for procalcitonin levels on the third day - larger concentrations of this marker were associated with death for the patient; on day 7 - weaker inverse correlation (p < 0.05, r -0.246), by the end of treatment - a significant inverse correlation at p < 0.001, r -0.393. A correlation between D-dimer and the outcome of the stay was revealed - on the 3rd day and at the end of treatment - in both cases the correlation is inverse, quite significant (p < 0.01, r-0.237and p < 0.001, r-0.512 respectively). Higher ferritin levels correlated with death when determined in the late period of hospitalization - inverse correlation at p < 0.001, r-0.447.
Markers as outcome predictors | Laboratory markers were measured daily. For correlation analysis, control days of measurements were chosen: days 1-3-7-15.
  According to the results of ROC analysis predictively significant for mortal outcome (*AUC values are close to 1.0, at the significance level P =0.05) were: procalcitonin level on days 3, 7 and 15, CRP level on days 7 and 15, levels of D-dimer on days 3, 7 and 15, ferritin on days 3 and 7

SECONDARY OUTCOMES:
the correlation between the level of biomarkers and the degree of infiltration of lung tissue | Laboratory markers were measured daily. For correlation analysis, control days of measurements were chosen: days 1-3-7-15.
  The correlation between the level of biomarkers and the degree of infiltration of lung tissue (CRP, D-dimer, ferritin at the beginning of treatment and at the end of treatment, procalcitonin at the end of treatment) was identified. This correlation was direct in all cases.
The level of D-dimer quite significantly negatively correlated with the duration of stay in the intensive care unit | Laboratory markers were measured daily. For correlation analysis, control days of measurements were chosen: days 1-3-7-15.
  The level of D-dimer quite significantly (p < .001) negatively correlated with the duration of stay in the intensive care unit when assessed on days 1, 3 and at the end of treatment, but such a correlation was not detected on day 7.
The inverse correlation was found for procalcitonin and the patient-bed-days in the intensive care unit | Laboratory markers were measured daily. For correlation analysis, control days of measurements were chosen: days 1-3-7-15.
  The inverse correlation was found for procalcitonin and the duration of patient's stay in the intensive care unit - on day 3 (p < .05) and at the end of treatment (p< .01).

CONTACTS AND LOCATIONS:
Overall Officials: Aissulu Issabekova, MD, Study Chair — Karaganda Medical University
Locations (1):
- Karaganda Medical University, Karaganda, Kazakhstan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT06460753/Prot_SAP_000.pdf